CLINICAL TRIAL: NCT00645047
Title: Veterans Telemedicine Outreach for PTSD Services
Acronym: VTOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: DHI 07-054
Record Dates: First submitted 2008-03-19; First posted 2008-03-27 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2016-11

CONDITIONS: PTSD
Keywords: PTSD; Telemedicine; Patient-Centered Care; Professional Patient Relationship; Psychotherapy; Cognitive Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine CBT (Experimental): Cognitive behaviour therapy (CBT) delivered using videoconference telemedicine.
  Interventions: Behavioral: Telemedicine CBT
- In-Person CBT (Active Comparator): Cognitive behaviour therapy (CBT) delivered using in-person consultation.
  Interventions: Behavioral: In-Person CBT

INTERVENTIONS:
Behavioral: Telemedicine CBT — Use of Videoconfrence Technology To Provide Cognitive Therapy
  Arms: Telemedicine CBT
Behavioral: In-Person CBT — In-Person Provision Of Cognitive Therapy
  Arms: In-Person CBT

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) is considered a major public health problem in the U.S. due to its high prevalence and high rates of disability associated with the disorder. For thousands of veterans, PTSD is a chronic disorder, resulting directly from military service that causes substantial psychological suffering and social disability. Barriers to PTSD care include poor access, mistrust, and lack of benefit from traditional treatments. This project addresses two very important and timely questions. First, can telemedicine be used as a tool to extend effective, specialized mental health services such as, cognitive processing therapy (CPT), to veterans with poor access to care? Second, does therapy delivered by telemedicine effect the quality of care in terms of clinical outcomes (PTSD severity, Quality of Life), and the quality of patient-therapist interaction (patient satisfaction & communication)? By answering these questions, this study will provide valuable knowledge for VA researchers, clinicians, and policy makers. The study findings will have direct implications related to making specific recommendations regarding telemedicine utilization to deliver specialized mental health services for veterans suffering from PTSD.

DETAILED DESCRIPTION:
Anticipated Impact on Veterans' Healthcare: This project addresses two very important and timely questions related to the VHA's mission to provide state of the art care to OEF and OIF veterans. First, can telemedicine be used as a tool to extend effective, specialized mental health services such as, cognitive processing therapy (CPT), to veterans with poor access to care? Second, does therapy delivered by telemedicine effect the quality of care in terms of clinical outcomes (PTSD severity, Quality of Life), and the quality of patient-therapist interaction (patient satisfaction & communication)? By answering these questions, this study will provide valuable knowledge for VA researchers, clinicians, and policy makers. The study findings will have direct implications related to making specific recommendations regarding telemedicine utilization to deliver specialized mental health services for veterans suffering from PTSD.

Project Background/Rationale: Post-Traumatic Stress Disorder (PTSD) is considered a major public health problem in the U.S. due to its high prevalence and high rates of disability associated with the disorder. For thousands of veterans, PTSD is a chronic disorder, resulting directly from military service that causes substantial psychological suffering and social disability. Barriers to PTSD care include poor access, mistrust, and lack of benefit from traditional treatments.

However, recently developed evidenced based treatments like CPT are very effective. Unfortunately, these treatments are not widely available, as a large proportion of veterans live in rural communities and have poor access to specialized mental health care. The VA hospital system currently supports sophisticated telemedicine technology that can provide CPT to veterans in their home communities. The proposed project will assess the quality of CPT provided via telemedicine and its impact on outcomes, and is therefore, directly related to the VA's mission to provide advanced, accessible, and high quality health care to all eligible veterans regardless of place of residence: "Right care in the right place, at the right time".

Project Objectives: The objective of the proposed study is to conduct a systematic comparison of PTSD outcomes for veterans receiving cognitive processing therapy via telemedicine vs. in-person care. The patient-therapist relationship is central in establishing an effective therapeutic relationship and is strongly influenced by communication. Consequently, this project will also compare provider-patient communication during telemedicine consultations vs. in-person consultations.

Project Methods: We propose a randomized clinical trial of 254 patients receiving cognitive processing therapy either via telemedicine or by in-person care. Telemedicine visits will occur at La Jolla VA in San Diego and in-person visits will occur at the Mission Valley VA Clinic in San Diego. Veterans with PTSD will be enrolled from the primary care and mental health clinics at the above sites. Clinical services will be provided by 10 participating providers with specialized training in CPT. Therapy will be provided over 12 weekly sessions lasting 60 minutes each. Previously validated and widely used measures of PTSD symptom severity (Clinician-Administered PTSD Scale, PTSD Checklist ) and health related quality of life (SF-36) will be measured at baseline, at completion of therapy, and at 6 months follow-up. In addition, we will measure and compare the quality of verbal and non-verbal patient-provider communication for in-person and telemedicine visits via video recordings of visits, which will be analyzed using the Roter Interaction Analyses System. Patient and provider satisfaction will be measured post therapy with previously validated questionnaires. Statistical methods will include descriptive analyses, reliability analyses, and hypothesis testing using linear mixed models.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of chronic PTSD due to combat; co-morbid mood and anxiety disorders are expected, and will be permitted (to maximize generalizability) if PTSD symptoms are judged to be predominant based on primacy and severity of symptoms; the proposed treatment often ameliorates depression and anxiety symptoms;
2. age 18 or older; and
3. English fluency.

Exclusion Criteria:

1. unmanaged dementia, psychosis or manic episodes in past year;
2. substance abuse or alcohol dependence in past year as measured by AUDIT;
3. concurrent psychotherapies targeting PTSD or depression (veterans who are engaged in treatment for non-PTSD symptoms, for example, 12-step programs for substance problems, will be eligible);
4. severe cardiovascular or respiratory disease that would make it difficult to ensure regular attendance at psychotherapy sessions;
5. severe impairments in speech, vision, or hearing; and
6. head trauma resulting in loss of consciousness longer than 20 minutes.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zia Agha, MD MS, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorp SR, Fidler J, Moreno L, Floto E, Agha Z. Lessons learned from studies of psychotherapy for posttraumatic stress disorder via video teleconferencing. Psychol Serv. 2012 May;9(2):197-9. doi: 10.1037/a0027057. PMID 22662733
- [Result] Backhaus A, Agha Z, Maglione ML, Repp A, Ross B, Zuest D, Rice-Thorp NM, Lohr J, Thorp SR. Videoconferencing psychotherapy: a systematic review. Psychol Serv. 2012 May;9(2):111-131. doi: 10.1037/a0027924. PMID 22662727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telemedicine CBT | In-Person CBT
Started | 103 | 104
Post | 74 | 80
Completed | 60 (6 month follow up) | 65
Not Completed | 43 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemedicine CBT | In-Person CBT | Total
Number analyzed (Participants) | 103 | 104 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (14.1) | 45.6 (13.5) | 48.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing Data
  Participants
    number analyzed (Participants) | 97 | 102 | 199
    Female | 19 | 26 | 45
    Male | 78 | 76 | 154
Region of Enrollment [Number; unit: participants]
  United States | 103 | 104 | 207

OUTCOME MEASURES:

1. Primary Outcome: CAPS - PTSD Symptom Severity Score
Description: The CAPS-5 is a 30-item clinician administered interview designed to diagnose current and lifetime PTSD and to assess PTSD symptom-severity over the past week. The interview assesses 20 DSM-5 PTSD symptoms as well as onset, duration, distress, and functional impact, overall validity, PTSD severity, and presence of dissociation. Prior to assessing symptoms, the clinical interviewer works with the patient to establish an index-trauma and each follow-up question focuses on symptoms as they relate to the index trauma.
  Severity Rating
  0. Absent; 1. Mild / subthreshold; 2. Moderate / threshold; 3. Severe / markedly elevated; and 4. Extreme / incapacitating.
  Higher scores means more severe symptoms. Total symptom severity score may range from 0-80, higher scores meaning more severe symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 103 | 104
units on a scale | 71.3 (17.8) | 72.5 (18.4)

2. Primary Outcome: CAPS - PTSD Symptom Severity Score
Description: as for outcome 1
Time Frame: Post Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 74 | 80
units on a scale | 62.1 (27.5) | 53.4 (26.2)

3. Primary Outcome: CAPS - PTSD Symptom Severity Score
Description: as for outcome 1
Time Frame: 6 Month Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 60 | 65
units on a scale | 56.6 (28.5) | 57.3 (26.9)

4. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
  Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Validity has been assessed against an independent structured mental health professional (MHP) interview. PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 103 | 104
units on a scale | 15.6 (6.5) | 16.4 (12.7)

5. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: as for outcome 4
Time Frame: Post Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 74 | 80
units on a scale | 12.9 (7.2) | 12.7 (6.7)

6. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: as for outcome 4
Time Frame: 6 Month Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 60 | 65
units on a scale | 12.5 (6.8) | 13.3 (6.9)

7. Secondary Outcome: PTSD Checklist (PCL)
Description: PTSD Checklist-Military Version (PCL). The PCL is a 17-item self-report measure of the 17 DSM-IV symptoms of PTSD. The PCL has a variety of purposes, including screening individuals for PTSD, diagnosing PTSD, and monitoring symptom change during and after treatment.
  A total symptom severity score (range = 17-85) can be obtained by summing the scores from each of the 17 items that have response options ranging from 1 "Not at all" to 5 "Extremely".
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 103 | 104
units on a scale | 59.1 (13.7) | 58.5 (12.6)

8. Secondary Outcome: PTSD Checklist (PCL)
Description: as for outcome 7
Time Frame: Post Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 74 | 80
units on a scale | 51.3 (16.3) | 49.3 (16.7)

9. Secondary Outcome: PTSD Checklist (PCL)
Description: as for outcome 7
Time Frame: 6 Month Visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telemedicine CBT | In-Person CBT
Number analyzed (Participants) | 60 | 65
units on a scale | 48.3 (17.0) | 51.5 (16.7)

ADVERSE EVENTS:
Time Frame: 1 month and 6 months
Arm/Group | Telemedicine CBT | In-Person CBT
Serious Adverse Events (participants affected / at risk) | 0/103 | 2/104
Other Adverse Events (participants affected / at risk) | 0/103 | 1/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telemedicine CBT (N=103) | In-Person CBT (N=104)
Heart arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
5150 Danger to self and others (Psychiatric disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telemedicine CBT (N=103) | In-Person CBT (N=104)
ER Visit (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days